CLINICAL TRIAL: NCT01423565
Title: Comparison of Constant Current to Constant Voltage Stimulation in Subthalamic DBS for Parkinson's Disease
Brief Title: Comparison of Constant Current to Constant Voltage Stimulation in Subthalamic Deep Brain Stimulation for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Israel Zvi, Dr. Zvi Israel, Director, Functional Neurosurgery, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 386150-HMO-CTIL
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; Parkinson's Disease; Subthalamic Nucleus; Constant Current
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental)
  Interventions: Device: Deep Brain Stimulation (Medtronic, Activa PC)

INTERVENTIONS:
Device: Deep Brain Stimulation (Medtronic, Activa PC) — Following subthalamic nucleus deep brain stimulation patients will be randomized to receive either constant current or constant voltage stimulation and subsequently "crossed over" to receive the other type of stimulation
  Other Names: Medtronic; Activa PC

SUMMARY:
HYPOTHESIS: Constant current stimulation for STN DBS will allow better and more stable control of Parkinson's disease symptoms than constant voltage stimulation.

Subthalamic nucleus (STN) deep brain stimulation (DBS) is an established therapy for advanced Parkinson's disease (PD). Two types of implantable pulse generators (IPGs) are available, differing on whether voltage or electrical current is controlled. Constant current IPGs provide a specific electrical current and will automatically adjust the voltage depending on the impedance, while the current applied by constant voltage IPGs will depend on the tissue impedance that may change over time. No study has compared the clinical differences of these two electronic modalities.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is an established therapy for neurological and psychiatric disorders, being one of the most important therapies in functional neurosurgery to date. Class I evidence shows that subthalamic nucleus stimulation (STN) for Parkinson's disease (PD) is more effective than the best medical therapy (1,2). Globus pallidus internus stimulation for primary dystonia has an improvement rate of up to 70%(4) and is considered the main surgical treatment for this pathology. Symptom improvement in essential tremor is well documented. Pain, epilepsy, psychiatric disorders such as Tourette syndrome, obsessive - compulsive disorder and depression are promising applications of DBS. Obesity, memory improvement, aggressiveness, drug addiction, minimal conscious state and hypertension are areas of continuing investigation as potential applications of DBS.

The clinical effects of DBS result from the delivery of electrical charge to brain tissue. The way this electrical charge is delivered depends on the electronics of implantable pulse generators (IPGs). IPGs apply pulses of electrical stimulation in which voltage or current increases from zero to a maximum value for a period of time (order of tens of microseconds) and then returns to zero.

There are two types IPGs , differing on whether voltage or electrical current is controlled (3).

1. Constant - voltage IPGs: in this type of IPG there is control over the maximum voltage associated with each pulse. The maximum current will vary depending on the impedance. A specific voltage is programmed. The amount of electrical current delivered with a constant voltage depends on the impedance of the tissue and the electrodes. Thus, the voltage will not indicate how much electrical current is given; the resistance will determine this parameter.
2. Constant - current IPGs: provide a specific electrical current and will automatically adjust the voltage depending on the impedance. The strength of stimulation will remain the same regardless of changes in the impedance. The difference in impedances on each electrode and the intersubject variability in impedances will not alter the electrical current by modifying the voltage.

Until fairly recently, only constant voltage IPG's have been available for use. A newer generation of IPG's have been available for more than a year that can provide either constant voltage or constant current according to physician and patient preference. There is no evidence yet to support the preferential use of one modality over the other.

IMPORTANCE OF THE STUDY Following DBS electrode implantation, the impedances within the same patient can vary widely. Surgical implantation changes tissue impedance, being usually higher immediately after surgery. In this case the patient will require higher electrical currents. After the initial tissue reaction subsides, the reduction of impedance will generate an increase of the charge density. For this reason it is commonplace to wait at least 2 weeks after electrode implantation before programming the IPG.

Furthermore, different contacts on the same DBS lead can have widely varying impedances. Effects or side effects associated with stimulation of one electrode contact often cannot be applied to a different contact on the same DBS lead in the same patient because the impedances may differ.

The range of impedances that can be measured will depend on the choice of voltage. In some patients, the voltage used therapeutically may not be enough to allow an accurate measure of the impedances, causing confusion regarding the structural and electrical integrity of the IPG.

For all the above mentioned factors, the clinical results in patients with constant - voltage IPGs will depend on the experience of the operator to deal with the different aspects related to tissue and electrode impedances to achieve the desired current. The electronic properties of constant - current IPGs allows the system to make voltage adjustments in order to maintain the desired current and the subsequent clinical effect. This has been the theoretical background for the development of constant current IPG's; whether or not this theory is true in practice is the subject of this study.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Subthalamic Deep Brain Stimulation Surgery

Exclusion Criteria:

* Any patient not meeting the inclusion criteria

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Impact of constant current on motor effects of STN DBS | 1 month
  To assess any clinical impact of changing the electronic modality of IPGs from constant - voltage to constant - current in patients with advanced PD after STN stimulation in terms of motor examination according to the Unified Parkinson's Disease Rating Scale (UPDRS) III.

SECONDARY OUTCOMES:
Impact of constant current on psychocognitive affective status | 1 month
  To assess the clinical impact of changing the electronic modality of IPGs from constant - voltage to constant - current in patients with advance PD after STN in terms of cognitive function, behavior, mood, quality of life and emotional processing according to the UPDRS I, UPDRS II, Hamilton Rating Scale for Depression (HAM-D17), Beck Depression Inventory (BDI), Clinical Global Inventory (CGI), Parkinson's disease questionnaire (PDQ-39), Addenbrooke's Cognitive Examination (ACE), Frontal Assessment Battery (FAB) and Hebrew version of the Montreal Affective Voices paradigm.

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Israel, MBBS, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel